CLINICAL TRIAL: NCT04699526
Title: Evaluation of Universal Prevention Curriculum for Schools in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HBSA (Other)
Responsible Party: Principal Investigator, Mallie J. Paschall, Ph.D., Senior Research Scientist, HBSA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Peru UPC Evaluation
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Received UPC training, school policy and climate interventions, and Unplugged prevention program
  Interventions: Other: Universal Prevention Curriculum Training for Schools
- Control (No Intervention): Only implemented Unplugged prevention program

INTERVENTIONS:
Other: Universal Prevention Curriculum Training for Schools — School administrators and teachers participated in UPC training and formed prevention leadership action teams
  Arms: Intervention

SUMMARY:
This randomized controlled trial was conducted to evaluate a universal prevention curriculum (UPC) training for Peruvian school administrators and teachers to reduce substance use among students. Twenty-eight schools were randomly assigned to intervention and control conditions (14 per condition). Substance use outcomes were assessed with repeated cross-sectional samples of students in 2018 and 2019. Multi-level analyses were conducted to assess intervention effects on students' substance use and related problems.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted to evaluate a universal prevention curriculum (UPC) training for Peruvian school administrators and teachers to reduce substance use among students. Twenty-eight schools were randomly assigned to intervention and control conditions (14 per condition). Prevention leadership action teams were formed at intervention schools to implement evidence-based school policies and positive school climate activities, and a classroom substance use prevention curriculum. Substance use outcomes were assessed with repeated cross-sectional samples of students in 2018 and 2019. Multi-level analyses were conducted to assess intervention effects on students' substance use and related problems.

ELIGIBILITY:
Inclusion Criteria:

* Students in participating schools aged 11 to 19

Exclusion Criteria:

* Not attending participating schools

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27012 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Cigarette smoking | 1 year
  Smoking cigarettes
Alcohol use | 1 year
  Drinking alcoholic beverages
Heavy drinking | 1 year
  Five or more consecutive alcoholic drinks
Marijuana use | 1 year
  Marijuana use
Other drug use | 1 year
  Use of inhalants, cocaine, PCB, hallucinogens
Problems | 1 year
  Problems related to substance use
Friends' substance use | 1 year
  Friends' use of tobacco, alcohol, marijuana and other drugs
Awareness of school policies | 1 year
  Awareness of school tobacco and alcohol policies
School bonding | 1 year
  School bonding

CONTACTS AND LOCATIONS:
Overall Officials: Mallie J Paschall, PhD, Principal Investigator — HBSA
Locations (1):
- Prevention Research Center, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be available to other researchers upon request after completion of the current study in December 2022.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after completion of the current study in December 2022, and will be available for five years afterwards.
Access Criteria: Data access information will be provided by the Principal Investigator.